CLINICAL TRIAL: NCT03208023
Title: RESIPI for Reducing Perioperative Major Adverse Cardiac Events: A Phase II Prospective Randomized Controlled Trial
Brief Title: RESIPI for Reducing Perioperative Major Adverse Cardiac Events
Acronym: RESIPI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Futility
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Cheetah Medical Inc. (Industry)
Responsible Party: Principal Investigator, Matthew McEvoy, Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 170601
Record Dates: First submitted 2017-06-30; First posted 2017-07-05 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Inotropy; Fluid Management; Cardiac Event; Perioperative Cardiac Risk; Vascular Resistance; Hemodynamic Monitoring; Hemodynamic Management; Fluid Responsiveness
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard intraoperative care- no interventions (Active Comparator): Standard intraoperative hemodynamic monitoring and treatment at Vanderbilt University Medical Center - No study interventions
  Interventions: Other: No intervention
- RESIPI (Experimental): Intraoperative implementation of RESIPI management strategy, a structured hemodynamic monitoring and treatment plan: RESIPI includes normalization of vascular resistance, correction of fluid responsiveness, and inotropy, and hemodynamic monitoring with the Starling SV (Cheetah Medical).
  Interventions: Procedure: RESIPI Management Strategy

INTERVENTIONS:
Procedure: RESIPI Management Strategy — a structured hemodynamic monitoring and treatment plan: RESIPI includes normalization of vascular resistance, correction of fluid responsiveness, and inotropy, and hemodynamic monitoring with the Starling SV (Cheetah Medical, Inc).
  Arms: RESIPI
Other: No intervention — No intervention
  Arms: Standard intraoperative care- no interventions

SUMMARY:
This study aims to evaluate the effect of a novel hemodynamic management and monitoring strategy for reducing cardiac bio marker elevations and major adverse cardiac events.

DETAILED DESCRIPTION:
Modest elevations in cardiac biomarkers in the immediate postoperative period are associated with significantly increased risk of morbidity and mortality. The RESIPI model of hemodynamic monitoring and management in the perioperative period takes into account the dynamic interplay of vascular resistance, inotropy, and fluid management. This study aims to evaluate the effect of a novel hemodynamic management and monitoring strategy for reducing cardiac bio marker elevations and major adverse cardiac events.

ELIGIBILITY:
Inclusion Criteria:

* Revised Cardiac Risk Index greater than or equal to 1, history of diastolic dysfunction, or age greater than 55 years.
* Surgery type: Major Abdominal Oncologic Surgery
* Planned surgery length greater than or equal to 90 minutes with planned in-patient stay of at least 2 days

Exclusion Criteria:

* Patients who are unstable by current American Heart Association/American College of Cardiology Clinical Practice Guidelines
* Patients with Chronic Kidney Disease Stage IV or V
* Urgent/emergent surgical interventions (e.g. Level 1 or 2 by VUMC VOR definitions)
* No signs of ischemia, congestive heart failure, or volume overload: Creatinine Clearance greater than 30

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
B-typer Natriuretic Peptide (BNP) | Post Op day 1
  Change in BNP (>250 ng/ml)
Troponin | Post Op day 1
  Change in troponin (>=0.04%)

SECONDARY OUTCOMES:
All-cause mortality | 30 days post op
Major cardiac events | 30 days post op
  Occurrence of major cardiac events (new arrhythmia, myocardial ischemia/infarction, congestive heart failure, or in-hospital cardiac arrest)
Hospital length of stay | Approximately 3-5 days
Readmission rate (Emergency room or hospital) | 30 days post operative
Return to operating room | 30 days post operative
Total hospital cost | 30 days post operative
Occurrence of significant medical events | 30 days post operative
  Occurrence of significant medical events (stroke, delirium, pneumonia, new oxygen requirement, need for re-intubation, acute kidney injury (KDIGO criteria), hyperglycemia (glucose >180)
Days at home in first 30 days | 30 days post operative

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D McEvoy, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No